CLINICAL TRIAL: NCT00005051
Title: Phase II Study of First-Line Therapy of Ovarian Cancer With Sequential Regimens: Cisplatin-Prolonged Oral Topotecan (C-PORT) Followed by Paclitaxel/Carboplatin (PC)
Brief Title: Combination Chemotherapy in Treating Patients With Advanced Ovarian Epithelial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000067644; NYU-9913; NCI-G00-1720
Record Dates: First submitted 2000-04-06; First posted 2003-01-27 (Estimated); Last update posted 2012-11-09 (Estimated); Status verified 2003-12

CONDITIONS: Ovarian Cancer
Keywords: stage I ovarian epithelial cancer; stage II ovarian epithelial cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Carboplatin; Cisplatin; Paclitaxel; Topotecan

INTERVENTIONS:
Drug: carboplatin
Drug: cisplatin
Drug: paclitaxel
Drug: topotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy in treating patients who have advanced ovarian epithelial cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the toxicity and tolerance of sequential therapy with prolonged
* Determine the response rate and time to progression in this patient
* Determine the relative pharmacokinetics of IV and prolonged oral administration of topotecan in the same patients and compare the pharmacodynamics of topo-1 inhibition when given by IV or oral route.

OUTLINE:

* Regimen A: Patients receive cisplatin IV over 60-90 minutes on day 1 of each course. Topotecan IV is administered continuously on days 1-14 of course 1. Oral topotecan is administered twice daily on days 1-14 for courses 2, 3, and 4. Treatment repeats every 28 days for 4 courses.
* Regimen B: After completion of regimen A, patients receive paclitaxel IV over 3 hours followed by carboplatin IV over 30 minutes on day 1. Treatment repeats every 21 days for 4 courses.

PROJECTED ACCRUAL: A total of 30 patients (15 per arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed advanced ovarian epithelial carcinoma, regardless of quantity of disease post-surgery

  * Stage IC, II, III, or IV

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* SGOT no greater than 3 times upper limit of normal
* Bilirubin no greater than 2.0 mg/dL
* No clinically significant hepatic disorder

Renal:

* Creatinine no greater than 1.5 mg/dL OR
* Creatinine clearance greater than 60 mL/min
* No clinically significant renal disorder

Cardiovascular:

* No clinically significant cardiovascular condition

Other:

* Normal GI function allowing reliable administration of oral medication
* No active infection requiring systemic medical therapy within past week
* No other clinically significant medical condition (e.g., endocrine/metabolic or autoimmune disorder)
* No other prior malignancy within the past 5 years except nonmelanoma skin cancer or carcinoma in situ of the cervix
* No dementia or altered mental status that would preclude consent
* Not pregnant
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy for ovarian epithelial carcinoma

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy for ovarian epithelial carcinoma

Surgery:

* See Disease Characteristics

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-08; Primary Completion 2003-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard S. Hochster, MD, Study Chair — NYU Langone Health
Locations (10):
- United States (10):
  - New York Hospital Medical Center of Queens, Fresh Meadows, New York
  - Saint Vincent Catholic Medical Center of New York, New York, New York
  - NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York
  - St. Luke's-Roosevelt Hospital Center - Roosevelt Division, New York, New York
  - New York Weill Cornell Cancer Center at Cornell University, New York, New York
  - Mount Sinai Medical Center, NY, New York, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University, New York, New York
  - Albert Einstein Clinical Cancer Center, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin